CLINICAL TRIAL: NCT00734396
Title: Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Allograft Rejection After Renal Transplantation
Brief Title: Mesenchymal Stem Cells and Subclinical Rejection
Acronym: Measure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, M.E. J. Reinders, MD, PhD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P08.119; NL21298.000.08
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Organ Transplantation
Keywords: Mesenchymal stem cells; Allograft rejection; Subclinical rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Mesenchymal stem cell infusion — MSC infusion: two doses of 1-2x106 MSCs per kilogram body weight, intravenously, 7 days apart.
  Other Names: Bone marrow derived mesenchymal stem cells.

SUMMARY:
The purpose of the study is to test the safety and feasibility of autologous mesenchymal stem cell therapy in HLA-DR mismatched patients with subclinical rejection and or an increase in IF?TA in the renal biopsy 4 weeks or 6 months after renal transplantation.

DETAILED DESCRIPTION:
Kidney transplantation has improved survival and quality of life for patients with end-stage organ failure. Despite dramatic improvements in short-term survival, long-term survival of renal allografts has changed little during the past decade. Recently, it has been demonstrated that chronic lesions originate already very early after transplantation and that subclinical rejection (SCR) in protocol biopsies is a risk factor for late graft loss. However the efficacy of high-dose corticosteroids and other therapies for the treatment of SCR have been shown to be inadequate. Thus, despite the availability of a range of available medications there remains a need for therapeutic alternatives because patients may not respond to existing therapeutic choices, they do not show an improvement of the fibrosis reaction or an effect on long term survival, or they may develop immunosuppression induced serious (sometimes fatal) side effects and toxicities.

In recent years it has become evident that bone marrow (BM) derived mesenchymal stem cells have potent immunomodulatory effects. MSCs are pluripotent cells that can differentiate into several mesenchymal tissues, including fibroblasts, osteoblasts, adipocytes and chondrocyte progenitors. MSCs have potent immunosuppressive effects on T and B cells in vitro and in animal models of chronic inflammation. Encouraging results have been obtained in patients with steroid resistant acute and severe Graft versus Host Disease (GvHD). The investigators hypothesize that infusion of MSCs may similarly provide a novel treatment option in the treatment of patients with allograft rejection with less side effects than existing immunosuppressive therapies.This study will evaluate the safety and feasibility of MSC therapy in renal recipients.

In total 15 de novo renal recipients of 2 HLA-DR mismatched living donors, men and women, 18-65 years of age, will be recruited from the renal transplant clinics of the LUMC. Only patients with SCR abd or an increase in IF/TA in the protocol biopsy 4 weeks or 6 months after transplantation will receive MSC infusions. MSCs from patients without SCR in their biopsy will be only used for feasibility and function studies (as described earlier). Subjects will receive two doses of 1 x 10.6 MSCs per kilogram body weight, intravenously, 7 days apart. The investigators will investigate safety of MSC therapy by assessing the rate of (serious) adverse events in the study population using the World Health Organization (WHO) criteria. Feasibility will be obtained by determining the number of expanded MSCs in relation to the amount of BM collected, number of passages required and time to reach study target doses.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to participate in the study and has signed the informed consent.
* Recipients of a first kidney graft from a living HLA-DR mismatched donor (2 HLA-DR mismatches).
* Subjects included in the study must have kidney biopsy proven SCR 4 weeks after transplantation.
* Patients must be on triple immunosuppressive therapy of prednisone, CsA or tacrolimus and MMF according to current protocol.
* Panel Reactive Antibodies (PRA) ≤ 5%.
* Patients must be able to adhere to the study visit schedule and protocol requirements.
* If female and of child-bearing age, subject must be non-pregnant, non-breastfeeding, and use adequate contraception.
* Patients must be able to give informed consent and the consent must be obtained prior to any study procedure.

Exclusion Criteria:

* Double organ transplant recipient.
* Acute clinical rejection after transplantation.
* Patients with evidence of active infection or abcesses before MSC infusion.
* Patients suffering from hepatic failure.
* Patients suffering from an active autoimmune disease.
* Patients who have had a previous BM transplant.
* A psychiatric, addictive or any disorder that compromises ability to give truly informed consent for participation in this study.
* Use of any investigational drug after transplantation.
* Documented HIV infection, active hepatitis B, hepatitis C or TB according to current transplantation inclusion criteria.
* Subjects who currently have an active opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus (CMV), Pneumocystis carinii (PCP), aspergillosis, histoplasmosis, or mycobacteria other than TB) after transplantation.
* Malignancy (including lymphoproliferative disease) within the past 2-5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence) according to current transplantation inclusion criteria.
* Known recent substance abuse (drug or alcohol).
* Contraindications to undergo a BM biopsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary 1 Safety: rate of (serious) adverse events in the study population 2 Feasibility: determination of the number of expanded MSCs in relation to the amount of BM collected, number of passages required and time to reach study target doses | 2 years

SECONDARY OUTCOMES:
Secondary endpoints: 1 Presence of late acute rejection (in the 6 month biopsy compared with the 4 week biopsy). 2 Sirius red staining for renal cortical matrix accumulation. 3 Immunologic response before and after MSC infusion. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Reinders, MD, PhD, Principal Investigator — LUMC
Locations (1):
- Leiden Universitary Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Reinders ME, de Fijter JW, Roelofs H, Bajema IM, de Vries DK, Schaapherder AF, Claas FH, van Miert PP, Roelen DL, van Kooten C, Fibbe WE, Rabelink TJ. Autologous bone marrow-derived mesenchymal stromal cells for the treatment of allograft rejection after renal transplantation: results of a phase I study. Stem Cells Transl Med. 2013 Feb;2(2):107-11. doi: 10.5966/sctm.2012-0114. Epub 2013 Jan 24. PMID 23349326